CLINICAL TRIAL: NCT01711567
Title: Switching to Tenofovir Disoproxil Fumarate vs. Continuing Entecavir in Chronic Hepatitis B Patients With Partial Virologic Response During Entecavir Therapy: STEEP Study
Brief Title: Tenofovir Disoproxil Fumarate vs. Entecavir in Chronic Hepatitis B Patients With Partial Virologic Response to Entecavir
Acronym: STEEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Hyung Joon Yim, Associate professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEEP study
Record Dates: First submitted 2012-10-17; First posted 2012-10-22 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; TENOFOVIR; ENTECAVIR; PARTIAL RESPONDER
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- entecavir (Active Comparator): standard drugs
  Interventions: Drug: entecavir
- tenofovir (Active Comparator): study drugs
  Interventions: Drug: tenofovir

INTERVENTIONS:
Drug: tenofovir — tenofovir 300 mg qd
  Other Names: tenofovir (viread)
  Arms: tenofovir
Drug: entecavir — entecavir 0.5 mg qd
  Other Names: entecavir(baraclude) 0.5 mg qd
  Arms: entecavir

SUMMARY:
Entecavir, a potent antiviral agent, has been widely used for treatment-naïve chronic hepatitis B patients. However, about 20% of patients showed partial virologic response after 2 year of entecavir therapy (33% in HBeAg positive, 10% in HBeAg negative patients). Tenofovir is a nucleotide analogue with more potent antiviral activity. In addition, there is no cross resistance between the two drugs. Therefore it is assumed that tenofovir would be effective in the treatment of chronic hepatitis B patients who shows partial virologic response (detectable HBV DNA by real time PCR after 12 months of treatment) despite treatment with entecavir. In this study, we will compare the efficacy of switching to tenofovir with continuing entecavir in patients who shows partial virologic response to entecavir.

DETAILED DESCRIPTION:
The number of patients needed was calculated using PASS 2008. We hypothesized that two-thirds (65%) of the patients receiving TDF, and one-fifth (20%) of the patients receiving ETV, would achieve virologic response. We also assumed a 15% drop-out rate; thus, 22 patients were needed in each group to achieve 80% power to demonstrate a difference between the groups with a 5% level of significance.

The primary efficacy end point will be analyzed on a per-protocol basis, including only those patients who had completed the treatment schedule of study. In contrast, the intention-to-treat analysis will include all randomized subjects, even those dropped-out from the study before 12 months, as cases of treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. CHB patients (positive HBsAg more than 6 months)
2. Age 19 years old
3. HBeAg positive or negative patients
4. Patients receiving entecavir 0.5 mg more than 12 months
5. Detectable HBV DNA by real time PCR (HBV > 60 IU/mL)
6. Compensated liver function (Child-Pugh-Turcotte score ≤7, prothrombin time 3 sec above ULN or INR ≤1.5, serum albumin >3 g/dL, total bilirubin <2.5 mg/dL, no history of variceal bleeding, diuretics or ascites requiring paracentesis, hepatic encephalopathy)

Exclusion Criteria:

1. History of treatment with nucleotide analogue other than 0.5 mg of ETV
2. Serum creatinine level > 1.5 mg/dL or creatinine clearance < 50 mL/min
3. Absolute neutrophil count ≤ 1000 cell/mL
4. Hemoglobin level ≤ 10 g/dL in men or ≤ 9 g/dL in women
5. Antiviral resistance mutations on rtT184, rtS202, or rtM250 + rtM204V/I
6. A positive antibody test for human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
7. Pregnancy or lactation
8. HCC (in cases where alfa-fetoprotein levels were over 100 ng/mL, abdominal computed tomography or magnetic resonance image was performed to exclude HCC)
9. Untreated malignancy other than HCC.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Virologic response rate at year 1 (12 months) (HBV DNA < 20 IU/mL) | up to the end of year 1 (12 months)

SECONDARY OUTCOMES:
-Degree of HBV DNA reduction, mean HBV DNA, biochemical and serologic response rates, resistance, and adverse events at year 1 | up to the end of year 1 (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Yim, M.D., Principal Investigator — Korea University
Locations (1):
- Korea University Ansan Hospital, Ansan, Gyeonggi-do, South Korea